CLINICAL TRIAL: NCT03136809
Title: A Treatment Continuation Study for Patients With Amyotrophic Lateral Sclerosis/Motor Neuron Disease Who Have Successfully Completed Study CMD-2016-001
Brief Title: ALS Treatment Extension Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Collaborative Medicinal Development Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMD-2017-001
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — copper (II) diacetyl-di(N(4)-methylthiosemicarbazone); Copper

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label treatment extension study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cu(II)ATSM (Experimental): Cu(II)ATSM administered once daily
  Interventions: Drug: Cu(II)ATSM

INTERVENTIONS:
Drug: Cu(II)ATSM — copper-containing synthetic small molecule
  Other Names: diacetylbis(N(4)-methylthiosemicarbazonato) copper(II)

SUMMARY:
Treatment extension study for ALS/MND patients who participated in phase 1 study CMD-2016-001, completed assessments following six 28-day cycles of treatment, and whom the Investigator considers would benefit from continued CuATSM treatment.

DETAILED DESCRIPTION:
Treatment extension study for ALS/MND patients who participated in phase 1 study CMD-2016-001, completed assessments following six 28-day cycles of treatment, and whom the Investigator considers would benefit from continued CuATSM treatment. The same safety assessments as in the CMD-2016-001 study will be conducted after each cycle of treatment and the same efficacy assessments as in the CMD-2016-001 study will be conducted after every 3 cycles of treatment. Treatment will continue until the first to occur of (1) Investigator considers the patient is no longer deriving benefit from CuATSM treatment, (2) patient develops dependence on mechanical ventilation where dependence is defined as being unable to lie flat (supine) without it, unable to sleep without it, or daytime use, or (3) the patient withdraws consent.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study-specific procedures and treatment
* Documented completion of protocol-specific assessments following completion of six 28-day treatment cycles in study CMD-2016-001
* Principal Investigator considers the patient would benefit from continued treatment with Cu(II)ATSM
* Not taking riluzole or on the same (or lower) dose used during the CMD-2016-001 study
* Adequate bone marrow reserve, renal and liver function
* Women and men with partners of childbearing potential must take effective contraception while on study treatment

Exclusion Criteria:

* Inability to swallow oral medications or presence of a gastrointestinal disorder (e.g.,malabsorption) deemed to jeopardize intestinal absorption of study drug
* Dependence on mechanical ventilation (invasive or non-invasive) for any part of day or night, where dependence is defined as being unable to lie flat (supine) without it, unable to sleep without it, or daytime use
* Dementia that may affect either outcome measures or patient understanding and/or compliance with study requirements and procedures
* Current use of strong inducers or inhibitors of CYPs 2C19 and 2D6

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Tolerance of extended treatment | 24 months
  safety

SECONDARY OUTCOMES:
Treatment-related change in disease severity by ALS Functional Rating Scale - Revised (ALSFRS-R) | 24 months
  efficacy
Treatment-related change in cognitive function by Edinburgh Cognitive and Behavioral Assessment (ECAS) score | 24 months
  efficacy
Treatment-related change in respiratory function by seated forced vital capacity (FVC) | 24 months
  efficacy
Treatment-related change in quality of life by ALSSQOL-R score | 24 months
  efficacy
Treatment-related change in respiratory function by sniff nasal pressure (SNP) test | 24 months
  efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Rowe, MD, Principal Investigator — Macquarie University
Locations (1):
- Macquarie University, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Plan to publish study results in a peer-reviewed journal